CLINICAL TRIAL: NCT06579417
Title: Advanced Restriction Imaging and Reconstruction Technology for Prostate MRI (ART-Pro)
Brief Title: ART-Pro: Clinical Trial Evaluating Biparametric MRI and Advanced, Quantitative Diffusion MRI for Detection of Prostate Cancer
Acronym: ART-Pro
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: GE Healthcare (Industry); University of California, San Francisco (Other); Massachusetts General Hospital (Other); Weill Medical College of Cornell University (Other); Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Tyler Seibert, Associate Professor, University of California, San Diego
Other Study IDs: 804875
Record Dates: First submitted 2024-08-20; First posted 2024-08-30 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Multiparametric MRI; Biparametric MRI; Restriction Spectrum Imaging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- ART-Pro-1
  Interventions: Diagnostic Test: RSI MRI

INTERVENTIONS:
Diagnostic Test: RSI MRI — In ART-Pro-1, patients receive standard of care mpMRI, with addition of the RSI sequence, and subsets of the patients' images are read separately by two expert radiologists at the center, one of whom is the standard of care radiologist (Reader 1). Three research reports are generated using: bpMRI only (Reader 1), mpMRI (Reader 1), and bpMRI + RSIrs (Reader 2). The clinical report is submitted by Reader 1. Patients' future prostate cancer management will be recorded and used to evaluate the performance of the MRI techniques being tested.

SUMMARY:
This is a multicenter, multinational trial to evaluate advanced MRI techniques for improved detection of clinically significant prostate cancer (csPCa). The study will enroll 500 participants at 5 clinical centers (100 participants per center). The current standard MRI technique for prostate cancer screening is multiparametric MRI (mpMRI), but two drawbacks include need for intravenous (IV) contrast and dependence on radiologist expertise. The investigators expect that the combination of two other techniques, biparametric MRI (bpMRI) and Restriction Spectrum Imaging restriction score (RSIrs), will help non-expert radiologists achieve similar performance to expert radiologists using bpMRI or mpMRI for detection of csPCa, while avoiding the drawbacks that are present when using mpMRI.

DETAILED DESCRIPTION:
ART-Pro will be conducted in two phases (ART-Pro-1 and ART-Pro-2) and will evaluate bpMRI, mpMRI, and RSIrs (an advanced quantitative diffusion technique), for detection of csPCa. ART-Pro-1 will evaluate these techniques prospectively, by having each patients' MRI exam read by 2 expert radiologists, both using different subsets of the images to evaluate the different techniques. ART-Pro-1 will additionally evaluate RSIrs as a stand-alone quantitative biomarker. ART-Pro-2 will evaluate these same techniques retrospectively using radiologists of varying experience levels (novice, basic, and expert), and findings will be evaluated against the expertly created dataset from ART-Pro-1. Patients will be followed after initial enrollment for the purpose of extracting relevant medical outcomes, such as biopsy results or surgery pathology.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Referred for mpMRI of the prostate for suspicion of prostate cancer
* MRI is conducted using the standardized ART-Pro acquisition protocol

Exclusion Criteria:

* Currently incarcerated
* Previous diagnosis of prostate cancer
* Active non-prostate tumor(s) in structures of the body near the prostate
* Previous prostate surgery
* History of hip implant
* Metal implants or implanted devices in the body or other criteria that are deemed to require deviation from the usual acquisition protocol or scanning procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for a multiparametric prostate MRI at any of the five participating sites, with a clinical suspicion of prostate cancer and that meet all the inclusion/exclusion criteria
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients diagnosed with a grade group ≥2 prostate cancer on biopsy | 6 months

SECONDARY OUTCOMES:
Proportion of patients undergoing a biopsy that reveals no cancer or only grade group 1 prostate cancer | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Seibert, MD, PhD, Principal Investigator — University of California, San Diego
Locations (5):
- United States (4):
  - University of California San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Weill Cornell Medical College, New York, New York
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Derived] Baxter MT, Conlin CC, Bagrodia A, Barrett T, Bartsch H, Brau A, Cooperberg M, Dale AM, Guidon A, Hahn ME, Harisinghani MG, Javier-DesLoges JF, Kamran SC, Kane CJ, Kuperman JM, Margolis DJA, Murphy PM, Nakrour N, Ohliger MA, Rakow-Penner R, Shabaik A, Simko JP, Tempany CM, Wehrli N, Woolen SA, Zou J, Seibert TM. Advanced Restriction Imaging and Reconstruction Technology for Prostate Magnetic Resonance Imaging (ART-Pro): A Study Protocol for a Multicenter, Multinational Trial Evaluating Biparametric Magnetic Resonance Imaging and Advanced, Quantitative Diffusion Magnetic Resonance Imaging for the Detection of Prostate Cancer. Eur Urol Open Sci. 2024 Dec 20;71:132-143. doi: 10.1016/j.euros.2024.12.003. eCollection 2025 Jan. PMID 39811103